CLINICAL TRIAL: NCT04148794
Title: The Development and Evaluation of the Efficacy for Echo-assisted Advanced Life Support Advanced Life Support (eALS)
Brief Title: The Development and Evaluation of the Efficacy for Echo-assisted Advanced Life Support Advanced Life Support
Acronym: eALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201812023RINA
Record Dates: First submitted 2019-10-27; First posted 2019-11-04 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Education of Ultrasound
Keywords: advanced life support; ultrasound; point-of-care ultrasound; echo-assisted advanced life support

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Participants who join the class of eALS
  Interventions: Behavioral: echo-assisted advanced life support

INTERVENTIONS:
Behavioral: echo-assisted advanced life support — Integrated point-of-care ultrasound skill in to the setting of resuscitation, and critical condition patients.
  Educate the participants to use these protocols and monitoring if there were improvement of patient's outcomes

SUMMARY:
The investigators conduct this project for integrating the point-of care ultrasound skill (POCUS) in to the American Heart Association (AHA) Advanced Cardiopulmonary Life Support (ACLS) guidelines and other critical conditions. Through lecture, head-on practice and scenario simulations, junior physicians who are the participants would be more familiar with the practice of POCUS in the settings of resuscitation and on the critical condition patients. The investigators aimed to increased the success rate of resuscitation and improve the outcomes of critical condition patients.

The investigators also try to make a template of ultrasound education in the board of emergency medicine and critical care medicine.

DETAILED DESCRIPTION:
Advanced life support (ALS) is an important training course for junior physicians to learn how to manage critical patients. Ultrasound is an indispensable and easily accessible tool in emergency departments and critical care settings. Current guidelines suggested that ultrasound could be an integral part of resuscitative medicine. However, structured training is needed for better efficacy of ultrasound use during clinical use. The aim of this project is to incorporate ultrasound into the ALS course, including common critical diseases, such as dyspnea, shock, major trauma and cardiac arrests. Junior physicians at the National Taiwan University Hospital will be enrolled in this study as participants. Through lectures and hand-on practice, the junior physicians could be familiar with managing critical patients with ultrasound assistance. This study will be lasted for two years. In the 1st year, the investigators will establish the echo-assisted ALS (eALS) training course, set up assessment modules and simulation scenarios. In the 2nd year, the investigators will provide the formal eALS training course for 4 to 6 times, analyze the data and establish on-line learning modules. In addition, the investigators will promote the eALS course to other hospitals and other countries.

This pioneer study can provide experience of eALS training course and contribute to current medical education. Moreover, it can improve decision-making process and quality of care of the participants. Furthermore, the integrated on-line learning programs can be used to lessen the maturation time of the participants and would provide them to other departments and hospitals to improve patients' care.

ELIGIBILITY:
Inclusion Criteria:

* all physicians or health care providers who are not well-experienced in the board of any kind of ultrasound

Exclusion Criteria:

* nil

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The improvement of performance of participant in the practicing of ultrasound | 32 weeks
  Compare the pre-lecture written test and a post-lecture written test results. There is also a hands-on examination after the lecture, to evaluate the participants skills, by using scoring sheets.

OTHER OUTCOMES:
Cardiac arrest patients ROSC rates | 32 weeks
  The rate of return of spontaneous circulation of cardiac arrest patients before and after the lecture
Length of stay (hours) in the emergency department | up to 32 weeks
  We proposed that the disposition of patient would be faster after the lecture. We would try to compare the length of stay (hours) in the ED before and after the lecture
diagnostic accuracy of the participants after training | 4 weeks
  sensitivity and specificity for acute chest pain and dyspnea, comparing with the final diagnosis. The final diagnosis was made by the retrospective chart review by the experts.

CONTACTS AND LOCATIONS:
Overall Officials: Department of Emergency medicine, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No